CLINICAL TRIAL: NCT03806283
Title: Angiotensin 2 Receptor (AT2R) Expression/Activation in Endothelial Cells in Preeclampsia
Brief Title: Mechanisms of Pregnancy Vascular Adaptations
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2025-1352; 5R01HL134779-02 (NIH); A532860 (Other: UW Madison); SMPH/OBSTET & GYNECOL/OBSTET (Other: UW Madison); Protocol Version 12/23/2025 (Other: UW Madison); 2018-1368 (Other: UW-Madison IRB)
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pre-Eclampsia; Vascular Diseases
MeSH Terms: conditions — Pre-Eclampsia; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — omental tissue (research surgical excision) placental tissue (standard of care clinical delivery)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 no Preeclampsia: Cohort 1: mothers with no diagnosis of preeclampsia during pregnancy Omental Biopsy and placental collection will be performed
  Interventions: Procedure: Omental Biopsy
- Cohort 2 mild or severe Preeclampsia: Cohort 2: mothers with diagnosis of mild or severe preeclampsia during pregnancy Omental Biopsy and placental collection will be performed
  Interventions: Procedure: Omental Biopsy

INTERVENTIONS:
Procedure: Omental Biopsy — The surgeon and clinical care team will conduct the c-section to deliver the baby and the placenta as clinically indicated. After delivery, during the closing procedures, the surgeon will indicate a time for a participating Ob/Gyn physician on the study team to collect the omental bio-specimen. Omentum is frequently excised or removed for clinical reasons during surgical procedures. Omentum has small blood vessels within it that have been used for evaluation of vascular functional changes in research. The investigators wish to isolate one to three vessels of 5 to 7 cm length. The surgeon will then close and the clinical care team will resume their standard of care activities.

SUMMARY:
The investigators will collect omental tissue (research surgical excision) and placental tissue (standard of care clinical delivery) from both preeclamptic and non-preeclamptic women during their c-section and use these samples to study the blood vessels, specifically the expression/activation of the AT2R.

DETAILED DESCRIPTION:
Trial Design: The study is a comparison of two cohorts, those with and without preeclampsia during pregnancy. The team plans to investigate role of FABP4, PFAS and AT2 in modulation of vascular function/dysfunction using vessels isolated from the omental biopsies. The investigators will examine evidence of fetal vascular dysfunction mediated by decreased expression of AT2 in preeclampsia using vessels isolated from the placentas.

Study Population: The study will include pregnant women. The pregnant women will participate in the omental tissue collection, placenta collection, and the medical record review.

The study is expects a maximum enrollment of 166 pregnant women. This is because 52 omental biopsies and 104 placentas are required to meet proposed statistical considerations. Participants have the option of providing just one or both of the specimens. There is a possibility as few as 52 participants could be enrolled and a maximum of 166 participants could be enrolled to meet this requirement. There is an additional 10 participants enrollment built into the enrollment number to allow for replacement of subjects based on lack of clinical data in some participants, failure of tissue viability and hence experiments, and thus a maximum of 166 (156+10) participants could be enrolled.

This required enrollment is divided into two cohorts based on the diagnosis of preeclampsia: specimens in which the woman was diagnosed with preeclampsia during her pregnancy, and 26 of each type of specimen in which the woman was not diagnosed with preeclampsia during her pregnancy. Additionally, each cohort will be divided into two groups based on gender of the fetus.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18 to 40 years old
* Singleton gestation between 28 weeks, 0 days and 41 weeks, 0 days gestational age at the time of consent
* Undergoing caesarean section, either planned or otherwise with or without trial of labor

Exclusion Criteria:

* Treatment of severe hypertension by antihypertensive or use of magnesium sulfate after the patient is hospitalized for the diagnosis of preeclampsia.
* Any major fetal structural anomalies or aneuploidies
* Undergoing cesarean section for placental abruption or bleeding complications.
* Singleton gestation not within 36 weeks, 0 days and 41 weeks, 0 days gestational age at the time of enrollment (delivery)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women with or without Preeclampsia who will be undergoing a C-section
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Quantify the vascular AT2R expression and vascular function in placental and omental vascular arteries in both preeclamptic and controlled pregnancies. | 1 year
  The researchers will measure the amount and distribution of vascular angiotensin II type 1 receptor (AT1R) and AT2R during normal human pregnancy and in preeclampsia. The researchers will assess if AT2R expression varies with severity of preeclampsia. Based on pilot data, the researchers expect decreased AT2R and increased AT1R protein levels in preeclamptic vs normotensive vessels.
To test if ex-vivo treatment of AT2R agonists reverses the endothelial dysfunction and improves vasoconstriction in the preeclamptic vessels. | 1 year
  The researchers will quantify vascular AT2R expression and vascular function in placental and omental arteries of preeclamptic vs normal pregnant women. Vascular function studies will also test if ex vivo treatment with AT2R agonist reverses endothelial dysfunction and vasoconstriction in preeclamptic vessels.
To test AT2R mediated mechanisms on endothelial derived hyperpolarizing factor, nitric oxide and prostacyclin pathway of vascular relaxation to examine AT2's role in vaso-relaxation and AT2R mediated vasoconstrictor pathway will be defined. | 1 year
  To test the AT2R-mediated mechanisms, endothelium-derived hyperpolarizing factor (EDHF), nitric oxide, and prostacyclin (PGI2) pathways of vascular relaxation and AT1R-mediated vasoconstrictor pathways will be determined. Also, the expression of endothelial nitric oxide synthase, its activity state, and signaling components of EDHF and PGI2 pathways, as well as nitrate/nitrite and PGI2 production and changes in membrane potential, will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Sathish Kumar, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UnityPoint Health-Meriter Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT03806283/ICF_001.pdf